CLINICAL TRIAL: NCT02142959
Title: A Randomized, Double-blind, Vehicle-controlled, Parallel-group Phase 2 Study of the Efficacy, Safety, and Pharmacokinetics of RTA 408 Lotion in the Treatment of Patients at Risk for Radiation Dermatitis
Brief Title: RTA 408 Lotion in Patients at Risk for Radiation Dermatitis - PRIMROSE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Collaborators: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: RTA 408-C-1306
Record Dates: First submitted 2014-05-16; First posted 2014-05-20 (Estimated); Results first posted 2023-05-06 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer
Keywords: RTA 408; RTA 408 Lotion; Breast cancer; Radiation therapy; Radiation dermatitis; Oxidative stress; Inflammation; omaveloxolone
MeSH Terms: conditions — Breast Neoplasms; Radiodermatitis; Inflammation | interventions — Radiotherapy, Conformal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- omaveloxolone (RTA 408) Lotion 0.5% (Experimental): Omaveloxolone Lotion at a fixed dose of 0.5% administered topically to the radiation area, twice daily for approximately 9 weeks (up to a maximum of 16 weeks)
  Interventions: Drug: Omaveloxolone Lotion 0.5%; Radiation: 3D conformal radiation therapy
- omaveloxolone (RTA 408) Lotion 3% (Experimental): Omaveloxolone Lotion at a fixed dose of 3% administered topically to the radiation area, twice daily for approximately 9 weeks (up to a maximum of 19 weeks)
  Interventions: Drug: Omaveloxolone Lotion 3%; Radiation: 3D conformal radiation therapy
- Vehicle Lotion (Placebo Comparator): Vehicle Lotion administered topically to the radiation area, twice daily for approximately 9 weeks (up to a maximum of 16 weeks)
  Interventions: Drug: Vehicle Lotion; Radiation: 3D conformal radiation therapy

INTERVENTIONS:
Drug: Omaveloxolone Lotion 0.5% — Omaveloxolone lotion 0.5% will be applied topically twice-daily, for up to 13 weeks, during the course of radiation therapy
  Other Names: RTA 408 Lotion 0.5%
  Arms: omaveloxolone (RTA 408) Lotion 0.5%
Drug: Omaveloxolone Lotion 3% — Omaveloxolone lotion 3% will be applied topically twice-daily, for up to 13 weeks, during the course of radiation therapy
  Other Names: RTA 408 Lotion 3%
  Arms: omaveloxolone (RTA 408) Lotion 3%
Drug: Vehicle Lotion — Lotion vehicle manufactured to mimic RTA 408 lotion will be applied topically twice-daily, for up to 13 weeks, during the course of radiation therapy
  Arms: Vehicle Lotion
Radiation: 3D conformal radiation therapy — 45 50.4 Gy in 1.8 Gy per day, in addition to 10 - 16 Gy boost or 46 - 50 Gy in 2 Gy per day, in addition to 10 - 16 Gy boost, at the physician's discretion

SUMMARY:
Radiation dermatitis is experienced by almost all patients (up to 95%) receiving radiation therapy for cancer. Radiation dermatitis can be a serious condition because, in addition to its direct physical complications and the resulting impact on overall quality of life, it can also be a dose-limiting toxicity requiring changes to the prescribed course of radiation therapy. The most common strategy employed in an attempt to prevent or minimize radiation dermatitis involves moisturization of the irradiated area, use of a mild soap to keep the area clean, and minimizing exposure to potential mechanical irritants, such as scratching and rough clothing. However, this strategy has been shown to lack clinically significant efficacy. Consequently, there is a clinical need for new treatments that are effective in protecting against radiotherapy-induced oxidative stress and the subsequent development of radiation dermatitis.

Based on data from previous studies in animals and humans, Reata believes that omaveloxolone (RTA 408) Lotion may effectively prevent and mitigate radiation dermatitis in oncology patients undergoing radiation therapy.

This randomized, double-blind, vehicle-controlled, parallel-group trial will study the efficacy, tolerability and safety of two concentrations of omaveloxolone (RTA 408) Lotion (3% and 0.5%) versus vehicle in patients with breast cancer for whom radiation therapy is recommended.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patients (18 to 75 years of age, inclusive);
2. Patients diagnosed with ductal carcinoma in situ or non-inflammatory breast adenocarcinoma who have been referred for post-operative radiotherapy and have had no prior radiation treatment to that breast;
3. Patients planning to undergo 3D conformal radiation therapy to the whole breast (as part of breast-conservation therapy / lumpectomy) or chest wall (as part of post-mastectomy irradiation), with or without treatment of regional lymph nodes (i.e., axillary, supraclavicular, or internal mammary), using one of the following treatment schedules:

   1. 45 - 50.4 Gy in 1.8 Gy per day, in addition to 10-16 Gy boost
   2. 46 - 50 Gy in 2 Gy per day, in addition to 10-16 Gy boost;
4. Patients who received breast-conservation therapy / lumpectomy must be receiving ≥ 107% of the total radiation dose (calculated from the total radiation dose including boost) to any portion of the breast, based on radiation inhomogeneity, and/or have a breast volume ≥ 1200 cc;

Exclusion Criteria:

1. Patients with Stage T4 or Stage IV breast cancer;
2. Patients with prior radiation therapy to the breast treated in this study;
3. Patients with type V or VI skin according to the Fitzpatrick scale;
4. Patients with bilateral breast cancer;
5. Patients receiving partial breast irradiation therapy;
6. Patients with uncontrolled diabetes (HbA1c > 11.0%, historical values within 6 months of screening are acceptable);
7. Patients with collagen vascular disease or vasculitis;
8. Patients with concurrent active malignancy other than adequately treated basal cell carcinoma of the skin or carcinoma in situ of the cervix;
9. Patients with active bacterial, fungal or viral skin infections;
10. Patients with known active hepatitis B or hepatitis C infection;
11. Patients who intend to use any other topical cream, lotion or preparation applied to the radiation treatment area;
12. Patients receiving concomitant chemotherapy during the course of the planned radiation treatment regimen. Patients are eligible if they are receiving sequential, neoadjuvant or adjuvant chemotherapy that is not anticipated to be delivered during the time course of the radiation treatment regimen.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2014-06-30 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (27):
- United States (27):
  - Ironwood Cancer and Research Centers, Mesa, Arizona
  - St. Joseph's Hospital and Medical Center, Phoenix, Arizona
  - Arizona Cancer Center, Scottsdale, Arizona
  - University of Colorado Hospital, Dept. of Radiation Oncology, Aurora, Colorado
  - Norwalk Hospital, Norwalk, Connecticut
  - Lakeland Regional Cancer Center, Lakeland, Florida
  - John B. Amos Cancer Center, Columbus, Georgia
  - St. Vincent Anderson Regional Hospital Cancer Center, Anderson, Indiana
  - Parkview Research Center, Fort Wayne, Indiana
  - Radiation Oncology Associates - Parkview Research Center, Fort Wayne, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Willis-Knighton Cancer Center, Shreveport, Louisiana
  - University of Nebraska Medical Center - Eppley Cancer Center, Omaha, Nebraska
  - CaroMont Health Comprehensive Cancer Center, Gastonia, North Carolina
  - Sanford Health, Bismarck, North Dakota
  - St. John Health System, Tulsa, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Hughes Cancer Center, East Stroudsburg, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - AnMed Health Cancer Center, Anderson, South Carolina
  - 21st Century Oncology - Carolina Regional Cancer Center, Myrtle Beach, South Carolina
  - Spartanburg Regional Medical Center - Gibbs Cancer Center, Spartanburg, South Carolina
  - Sanford Research/USD, Sioux Falls, South Dakota
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Cancer Care Northwest, Spokane, Washington
  - Mayo Clinic - LaCrosse, La Crosse, Wisconsin
  - Columbia St. Mary's, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Omaveloxolone (RTA 408) Lotion 0.5% | Omaveloxolone (RTA 408) Lotion 3% | Vehicle Lotion
Started | 64 | 62 | 61
Completed | 59 | 59 | 55
Not Completed | 5 | 3 | 6
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 0 | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1 | 3
Not completed — Administrative Reasons | 1 | 0 | 1
Not completed — Missing | 0 | 1 | 0
Not completed — Treatment changed from radiation treatment to chemo | 0 | 0 | 1
Not completed — Patient didn't complete end of study visit | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat population (all randomized patients whether or not they received study drug)
Groups:
- Total: Total of all reporting groups
Arm/Group | Omaveloxolone (RTA 408) Lotion 0.5% | Omaveloxolone (RTA 408) Lotion 3% | Vehicle Lotion | Total
Number analyzed (Participants) | 64 | 62 | 61 | 187
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.7 (8.8) | 56 (10.2) | 56.6 (10.3) | 56.8 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 64 | 62 | 61 | 187
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 5 | 11
  Not Hispanic or Latino | 61 | 58 | 56 | 175
  Unknown or Not Reported | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 13 | 6 | 5 | 24
  White | 50 | 54 | 51 | 155
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 2 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 64 | 62 | 61 | 187

OUTCOME MEASURES:

1. Primary Outcome: Time-averaged Effect on Radiation Dermatitis Grade Measured With Common Terminology Criteria for Adverse Events (CTCAE, v 4.03) Following 3D Conformal Radiation Therapy to the Breast Following Topical Application of Omaveloxolone Lotion or Lotion Vehicle
Description: CTCAE Radiation dermatitis scoring:
  Grade 0 = No radiation dermatitis; Grade 1 = Faint erythema or dry desquamation; Grade 2 = Moderate to brisk erythema, patchy moist desquamation, mostly confined to skin folds and creases, moderate edema; Grade 3 = Moist desquamation in areas other than skin folds and creases, bleeding induced by minor trauma or abrasion; Grade 4 = Life-threatening consequences, skin necrosis or ulceration of full thickness dermis, spontaneous bleeding from involved site, skin graft indicated; Grade 5 = Death
Time Frame: Day 1 of radiation treatment through the last day of radiation treatment (maximum of 19 weeks), time averaged effect on radiation dermatitis reported
Population: Intent-to-treat population (all randomized patients whether or not they received study drug)
Measure: Least Squares Mean (95% Confidence Interval); unit: Grade
Arm/Group | Omaveloxolone (RTA 408) Lotion 0.5% | Omaveloxolone (RTA 408) Lotion 3% | Vehicle Lotion
Number analyzed (Participants) | 64 | 62 | 61
Grade | 1.1 [1.0 to 1.2] | 1.2 [1.1 to 1.3] | 1.2 [1.1 to 1.3]
Statistical Analysis 1: Comparison: Omaveloxolone (RTA 408) Lotion 0.5% vs Omaveloxolone (RTA 408) Lotion 3% vs Vehicle Lotion; Comparison of omaveloxolone lotion pooled (0.5% and 3%) versus vehicle lotion; Test type: Superiority; p = 0.237, Mixed Models Analysis — Omaveloxolone treatment arms were compared with Vehicle Lotion using a hierarchical testing strategy to control the overall type I error; Fixed factors: treatment grp & wk of visit; covariates of site, smoking status & surgery. Missing data imputed using each patient's worst-observation; LS Mean Difference Final Values = -0.1, 65% CI 2-sided [-0.2 to 0.0]
Statistical Analysis 2: Comparison: Omaveloxolone (RTA 408) Lotion 0.5% vs Vehicle Lotion; Comparison of Omaveloxolone Lotion 0.5% versus Vehicle Lotion; Test type: Superiority; p > 0.05, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; Fixed factor: treatment grp & visit wk; Covariates: site, smoking status & breast surgery. Missing data imputed using each patient's worst-observation; LS Mean Difference Final Values = -0.1, 95% CI 2-sided [-0.2 to 0.0]
Statistical Analysis 3: Comparison: Omaveloxolone (RTA 408) Lotion 3% vs Vehicle Lotion; Comparison of Omaveloxolone Lotion 3% versus Vehicle Lotion; Test type: Superiority; p > 0.05, Mixed Models Analysis; [statistical method as in outcome 1, analysis 2]; LS Mean Difference Final Values = 0, 95% CI 2-sided [-0.1 to 0.1]

ADVERSE EVENTS:
Arm/Group | Omaveloxolone (RTA 408) Lotion 0.5% | Omaveloxolone (RTA 408) Lotion 3% | Vehicle Lotion
All-Cause Mortality (participants affected / at risk) | 0/64 | 1/62 | 0/61
Serious Adverse Events (participants affected / at risk) | 4/64 | 3/62 | 0/61
Other Adverse Events (participants affected / at risk) | 49/64 | 54/62 | 50/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omaveloxolone (RTA 408) Lotion 0.5% (N=64) | Omaveloxolone (RTA 408) Lotion 3% (N=62) | Vehicle Lotion (N=61)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Incision site cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Omaveloxolone (RTA 408) Lotion 0.5% (N=64) | Omaveloxolone (RTA 408) Lotion 3% (N=62) | Vehicle Lotion (N=61)
Constipation (Gastrointestinal disorders) | 3 (3) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 3 (4)
Nausea (Gastrointestinal disorders) | 5 (5) | 3 (4) | 5 (5)
Asthenia (General disorders) | 0 (0) | 0 (0) | 2 (2)
Axillary pain (General disorders) | 3 (3) | 1 (1) | 0 (0)
Fatigue (General disorders) | 27 (29) | 27 (27) | 26 (28)
Pain (General disorders) | 3 (3) | 2 (2) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 2 (2) | 2 (2)
Breast infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 3 (3) | 0 (0)
Folliculitis (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 1 (1) | 2 (2)
Urinary tract infection (Infections and infestations) | 2 (2) | 2 (2) | 2 (2)
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) | 3 (3) | 1 (1)
Seroma (Injury, poisoning and procedural complications) | 2 (2) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 3 (4)
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 2 (2) | 3 (3) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 2 (2) | 4 (5)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Sciatica (Nervous system disorders) | 2 (2) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 3 (4) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 1 (1) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 2 (2) | 2 (2)
Breast pain (Reproductive system and breast disorders) | 20 (28) | 19 (27) | 18 (22)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (4) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 3 (3) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 2 (2)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 20 (22) | 17 (19) | 12 (12)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 1 (1)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (3) | 1 (2)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 19 (20) | 15 (15) | 18 (19)
Hot flush (Vascular disorders) | 3 (3) | 4 (4) | 4 (4)
Lymphoedema (Vascular disorders) | 1 (1) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2014-10-17): https://cdn.clinicaltrials.gov/large-docs/59/NCT02142959/Prot_000.pdf
  • Statistical Analysis Plan (2015-04-29): https://cdn.clinicaltrials.gov/large-docs/59/NCT02142959/SAP_001.pdf